CLINICAL TRIAL: NCT04847973
Title: Food As Medicine for Heart Failure
Acronym: FAM-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: Community Servings (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00001214
Record Dates: First submitted 2021-04-07; First posted 2021-04-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Heart Failure; Malnutrition
Keywords: heart failure; malnutrition; weight loss; cachexia; nutrition
MeSH Terms: conditions — Heart Failure; Malnutrition; Weight Loss; Cachexia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 12 weeks of medically-tailored meals (MTMs) (Experimental): 12 weeks of home-delivered medically-tailored meals (MTMs), prepared and delivered by the non-profit Community Servings. The MTM has be developed specifically for patients with heart failure, with an approximate protein intake range of 1.1-1.5 g/kg body weight/day and a maximum of 2000 mg sodium/day.
  Interventions: Other: Medically-Tailored Meals (MTMs)
- 12 weeks of protein supplementation shakes (Experimental): Participants will receive 1 bottle of Ensure Max Protein shake every day (any flavor option without caffeine, daily for 12 weeks) to take in addition to their standard diet, without MTM delivery.
  Interventions: Dietary Supplement: Protein supplementation shakes

INTERVENTIONS:
Other: Medically-Tailored Meals (MTMs) — 12 weeks of home-delivered MTMs, delivered weekly, containing food for 3 meals per day on 5 days of the week
  Arms: 12 weeks of medically-tailored meals (MTMs)
Dietary Supplement: Protein supplementation shakes — 12 weeks of 1 bottle of Ensure Max Protein shake every day, in addition to partcipants' standard diet
  Arms: 12 weeks of protein supplementation shakes

SUMMARY:
Malnutrition and unintentional weight loss are highly prevalent among patients with heart failure (HF), with approximately 50% of patients with heart failure meeting malnutrition criteria. Poor dietary quality and micronutrient deficiencies are associated with higher rates of HF hospitalization and mortality. Therefore nutritional interventions to improve dietary quality and prevent malnutrition development may represent an effective strategy to improve HF-related health status and survival outcomes. To date, there are no large clinical trials investigating the efficacy of 'food as medicine' to improve morbidity and mortality for patients with heart failure with reduced ejection fraction (HFrEF). The investigators plan to conduct a single-center, randomized pilot trial to assess the tolerability, feasibility, and efficacy of providing medically-tailored meals (MTMs) or protein supplementation shakes to patients with HFrEF and malnutrition. The investigators hypothesize that home delivery of MTMs or protein supplementation shakes will be feasible, well-tolerated and achieve a high degree of satisfaction for patients with HFrEF. The current pilot phase is a single arm non-randomized study. An initial phase has delivered a 12-week MTM dietary intervention. The MTMs are designed, prepared and delivered by our community based organized partner, Community Servings. A second phase will deliver a 12-week protein supplementation shake intervention, with 1 bottle to be consumed daily in addition to the participants' standard home diet. The investigators will measure HF-related health status, functional capacity, and biomarkers of heart failure and nutritional status before and after each study phase. The proposed study will facilitate a larger future randomized trial of nutritional intervention for patients with HFrEF and malnutrition, powered to examine the impact on HF hospitalizations and mortality.

DETAILED DESCRIPTION:
We plan to conduct a single-center pilot trial to assess the tolerability, feasibility, and efficacy of providing medically-tailored meals to patients with heart failure with reduced ejection fraction and malnutrition. We hypothesize that a nutritionally complete meal plan, targeting 1.1-1.5 g/kg/day protein intake, will improve symptomatology, functional capacity, and serum biomarkers of heart failure in this patient population. We have two primary objectives for this pilot study: 1) confirm tolerability, feasibility, and efficacy of prescribing MTMs or oral protein supplementation and 2) measure changes in functional capacity, patient-reported health status, and biomarkers of nutritional status and heart failure over the course of the study period. For this proposed study, we will test the following elements of this central hypothesis with 2 aims:

Aim 1 Tolerability, feasibility, and efficacy of prescribing medically-tailored meals or protein supplementation: Tolerability will be assessed with the validated 28-item dietary satisfaction score (DSat-28). Efficacy will be assessed by improvement in patient-reported health status questionnaires and feasibility will be assessed by the macronutrient intakes achieved on facilitated food recalls.

Aim 2 Functional capacity and serum biomarkers of nutrition/heart failure: Determine whether medically tailored meals improve symptomatology, functional capacity, and serum biomarkers of nutrition and heart failure in patients with advanced heart failure.

ELIGIBILITY:
Inclusion Criteria:

1. Systolic heart failure (left ventricular ejection fraction </=40%), with New York Heart Association (NYHA) class II-III symptoms
2. At least one prior hospitalization in the preceding 12 months
3. Evidence of malnutrition on the Short Nutritional Assessment Questionnaire (SNAQ) screening tool for malnutrition (score of 2 or more)
4. Have a fixed address within the Metro Boston region and availability of home refrigeration to accommodate the MTM deliveries
5. Able and willing to sign study consent
6. 18 years or above
7. Not currently pregnant and not imminently planning a pregnancy

Exclusion Criteria:

1. Prior heart transplantation or implantation of a left ventricular assist device
2. Patients with a non-cardiac etiology for a skeletal muscle disorder e.g. muscular dystrophy, cancer
3. Currently pregnant or planning to become pregnant
4. Food allergy, aversion, or dietary preference that cannot be accommodated by Community Servings
5. Systolic blood pressure at screening <90 mmHg, or heart rate >110 bpm
6. Galactosemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Kansas City Cardiomyopathy Questionnaire (KCCQ) | Change from start to end of 12-week MTM period
  Patient reported health measure (scale 0 to 100, higher indicates better health status)
Handgrip strength measurement in kg | Change from start to end of 12-week MTM period
  Upper extremity strength measured by dynamometer (higher kg achieved indicates greater strength)
Sit-to-stand test | Change from start to end of 12-week MTM period
  Lower extremity strength measure (lower time indicates greater strength)
6 minute walk test | Change from start to end of 12-week MTM period
  Strength and endurance measure
Diet Satisfaction scale (DSat-28) | Change from start to end of 12-week MTM period
  Dietary satisfaction measure

SECONDARY OUTCOMES:
Short Nutritional Assessment Questionnaire (SNAQ) | Change from start to end of 12-week MTM period
  Appetite questionnaire (score ranges 0 to 7, >/=3 indicating a severe malnutrition risk)
Facilitated food recall | Change from start to end of 12-week MTM period
  3-day 24-hour facilitated food recall
Weight | Change from start to end of 12-week MTM period
  Subject's body weight, measured on standing scale

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Vest, MBBS MPH, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No